CLINICAL TRIAL: NCT01478347
Title: A Phase 3b, Single-Center, Open-label Study to Assess the Safety of Novartis Meningococcal B Recombinant Vaccine When Administered at a 0, 2-Month Schedule in Healthy At-risk Adults
Brief Title: A Phase 3b Study to Assess the Safety of Novartis Meningococcal B Recombinant Vaccine When Administered in Healthy At-risk Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V72_37
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Neisseria, Meningitis, Group B, Vaccine, At-risk, Adults
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rMenB+OMV NZ (Experimental): Healthy adults (≥18 to ≤65 years), at high risk for meningococcal B disease due to routine occupational exposure to N. Meningitidis cultures (e.g. lab workers), were administered two injections of Recombinant meningococcal B (rMenB) + Outer Membrane Vesicle (OMV NZ) vaccine, 2 months apart, in part I of the study, were enrolled for optional blood draws and safety follow-up in part II of the study.
  Interventions: Biological: Recombinant meningococcal B + OMV NZ

INTERVENTIONS:
Biological: Recombinant meningococcal B + OMV NZ — 2 injections 2 months apart

SUMMARY:
The proposed study will evaluate the safety of the rMenB+OMV NZ in an adult population potentially at risk for meningococcal disease (e.g. lab workers).

In the second part of the study additional blood samples of high responding vaccinated subjects will be collected for the purpose of generating a control serum panel for the human serum bactericidal assay (hSBA) tests.

ELIGIBILITY:
Inclusion criteria:

1. 18 - 65 years of age inclusive who have given written informed consent at the time of enrollment;
2. Able to comprehend and follow all required study procedures;
3. Who are available for all the visits scheduled in the study (i.e., not planning to leave the area before the end of the study period);
4. In good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator;
5. Who were or might be routinely exposed to N. meningitidis cultures

Inclusion criteria for protocol part 2

1. 18 - 65 years of age inclusive;
2. At least 50 kg weight;
3. Blood pressure within the following ranges: Systolic 110-180; Diastolic 60-100;
4. Regular pulse rate (50-90 beats per minute) - exceptions are acceptable upon investigator's judgment;
5. Hematocrit higher than: 32% for women and 35% for males;
6. Visit 3 sera suitable as control for standardization of the SBA as confirmed by the central laboratory.

Exclusion criteria:

1. History of any serogroup B meningococcal vaccine administration
2. History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component;
3. Pregnancy or nursing (breastfeeding) mothers;
4. Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study. Oral, injected or implanted hormonal contraceptive, barrier methods (condom or diaphragm with spermicide), intrauterine device, surgical sterilization, transdermal delivery, congenital sterility or sexual abstinence are considered acceptable forms of birth control. If sexually active the subject must have been using one of the accepted birth control methods at least one months prior to study entry;
5. Known or suspected autoimmune disease or impairment/alteration of the immune system resulting from (for example):
6. Receipt of any chronic immunosuppressive therapy
7. Receipt of any chronic immunostimulants
8. Immune deficiency disorder, or known HIV infection
9. Known bleeding diathesis or any condition that may be associated with a prolonged bleeding time.
10. History or any illness/condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or pose additional risk to the subjects due to participation in the study.
11. Any significant chronic infection.
12. Any serious chronic or progressive disease according to judgment of the investigator (e.g. neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).

Exclusion criteria for protocol part 2:

1. Known or suspected autoimmune disease;
2. Any serious chronic or progressive disease according to judgment of the investigator (e.g. neoplasm, diabetes, cardiovascular, renal, hepatic, immunological, metabolic, urogenital, hematological, gastrointestinal, central nervous system disease);
3. Known bleeding diathesis or any condition that may be associated with a prolonged bleeding time;
4. History of fainting or seizure episodes;
5. Pregnancy
6. Any significant chronic infection;
7. Significant acute infections within the previous 2 weeks;
8. Known or suspected autoimmune disease or impairment/alteration of the immune system resulting from (for example):

   Receipt of any chronic immunosuppressive therapy; Receipt of any chronic immunostimulants; Immune deficiency disorder, or known HIV infection;
9. Significant acute illness within the previous 7 days or body temperature 38.0 C within the previous 3 days;
10. Receipt of systemic antibiotics within the previous 3 days (72 hours).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- UOC Medicina Interna 2, Azienda Ospedaliera Universitaria Senese, Siena, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a single center.
Pre-assignment Details: All enrolled subjects participated in the study.
Groups:
- rMenB+OMV NZ: Healthy adults (≥18 to ≤65 years), at high risk for meningococcal B disease due to routine occupational exposure to N. Meningitidis cultures (e.g. lab workers), were administered two injections of Recombinant Meningococcal B Vaccine with Outer Membrane Vesicle from the New Zealand Strain (rMenB + OMV NZ vaccine), 2 months apart, in part I of the study. In part II of the study subjects were re-enrolled for optional blood draws and safety follow-up.
Period: Visit 1-Visit 3 (Day 0-91) - Part I
Arm/Group | rMenB+OMV NZ
Started | 18
Completed | 17
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Visit 4-Visit 7 (Day 151-331) - Part II
Arm/Group | rMenB+OMV NZ
Started | 12
Completed | 4
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Healthy adults (≥18 to ≤65 years), at high risk for meningococcal B disease due to routine occupational exposure to N. Meningitidis cultures, were administered two injections of rMenB + OMV NZ vaccine, 2 months apart in part I (Visit 1-Visit 3). In part II (Visit 4-Visit 7), subjects were re-enrolled for optional blood draws and safety follow-up.
Groups:
- rMenB+OMV NZ: Healthy adults (≥18 to ≤65 years), at high risk for meningococcal B disease due to routine occupational exposure to N. Meningitidis cultures (e.g. lab workers), were administered two injections of rMenB + OMV NZ vaccine, 2 months apart, in part I of the study. 18 subjects were enrolled in part I of the study.
  In part II of the study, subjects were re-enrolled for optional blood draws and safety follow-up. Of the 18 subjects enrolled in part I of the study, only 12 subjects continued participation into protocol part II of the study. Only 11 subjects (one subject was withdrawn after visit 3 due to "lost to follow-up) were included in the safety set and therefore contributed to the baseline characteristics data.
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 18
Age, Customized [Mean (Standard Deviation); unit: years] — Of the 18 subjects enrolled for part I of the study, only 12 subjects continued participation into protocol part II of the study. Of these, 11 subjects were included in safety set.
  years
    rMenB (part I; N=18) | 34.5 (5.7)
    rMenB (part II; N=11) | 34.1 (5.6)
Sex/Gender, Customized [Number; unit: subjects]
  rMenB( part I; female) | 13
  rMenB( part I; male) | 5
  rMenB( part II; female) | 8
  rMenB( part II; male) | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events, Following Vaccination With Two Injections of rMenB+OMV NZ Vaccine Between Day 1 Through Day 91.
Description: The number of subjects with serious adverse events (SAE), medically attended adverse events and adverse events (AEs) leading to premature withdrawal, following two injections of rMenB+OMV NZ vaccine are reported.
Time Frame: Day 1 to day 91
Population: This analysis was done on the safety set population i.e all subjects in the exposed set with unsolicited adverse event data for part one of the study.
Measure: Number; unit: subjects
Groups:
- rMenB+OMV NZ: Healthy adults (≥18 to ≤65 years), at high risk for meningococcal B disease due to routine occupational exposure to N. Meningitidis cultures (e.g. lab workers), were administered two injections of rMenB + OMV NZ vaccine, 2 months apart, in part I of the study. In part II of the study subjects were re-enrolled for optional blood draws and safety follow-up.
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 18
subjects
  Medically attended AEs | 2
  At least possibly related medically | 0
  SAEs | 0
  At least possibly related SAEs | 0
  Premature withdrawals due to AEs | 0

2. Primary Outcome: Number of Subjects (Who Had Received Two Injections of rMenB+OMV NZ Vaccine in Part I of This Study) Reporting Unsolicited Adverse Events During Safety Follow-up (Part II of the Study).
Description: The number of subjects (who had received two injections of rMenB + OMV NZ vaccine in the part I of this study) reporting unsolicited AEs during the safety follow-up in part II of the study, are reported. Unsolicited AEs in part two of the study include - AEs considered to be related to blood draw procedure and all SAEs.
Time Frame: Day 92 to day 331
Population: This analysis was done on the safety set population i.e all subjects in the exposed set with unsolicited adverse event data for part two of the study.
Measure: Number; unit: subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 11
subjects
  All AEs | 0
  SAEs | 0
  At least possibly related SAEs | 0

ADVERSE EVENTS:
Time Frame: All serious adverse events and other unsolicited adverse events collected from Day 1 to Day 331 (throughout the study) for subjects who participated in both part I and II of the study, are reported.
Arm/Group | rMenB+OMV NZ
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB+OMV NZ (N=18)
Pharyngitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement: the terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial